CLINICAL TRIAL: NCT00003117
Title: Single-Agent Versus Combination Chemotherapy in Advanced NSCLC: A CALGB Randomized Trial of Efficacy, Quality of Life, and Cost-Effectiveness
Brief Title: Paclitaxel With or Without Carboplatin in Treating Patients With Advanced Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-9730; U10CA031946 (NIH); CLB-9730; CDR0000065871 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 1999-11-01; First posted 2004-05-19 (Estimated); Last update posted 2016-06-30 (Estimated); Status verified 2016-06

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; squamous cell lung cancer; large cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; adenocarcinoma of the lung; adenosquamous cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung | interventions — Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Paclitaxel (Experimental): Patients receive paclitaxel IV over 3 hours on day 1 of each course. Treatment is repeated every 21 days for 6 courses in the absence of tumor progression or unacceptable toxicity. Quality of life assessments are conducted before treatment and at 2, 6, 9, and 12 months. Patients are followed every 3 months for 2 years, then every 6 months until disease progression or death.
  Interventions: Drug: paclitaxel
- Paclitaxel + Carboplatin (Experimental): Patients receives paclitaxel as in Arm I, followed by carboplatin IV over 1 hour. Treatment is repeated every 21 days for 6 courses in the absence of tumor progression or unacceptable toxicity. Quality of life assessments are conducted before treatment and at 2, 6, 9, and 12 months. Patients are followed every 3 months for 2 years, then every 6 months until disease progression or death.
  Interventions: Drug: carboplatin; Drug: paclitaxel

INTERVENTIONS:
Drug: carboplatin
  Arms: Paclitaxel + Carboplatin
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Randomized phase III trial to compare the effectiveness of paclitaxel with or without carboplatin in treating patients who have recurrent, stage IIIB, or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the overall survival of patients with non-small cell lung cancer treated with paclitaxel alone or in combination with carboplatin. II. Compare the quality of life of these patients treated with these chemotherapy regimens. III. Compare the response rates and the toxic effects of the two regimens in this patient population.

OUTLINE: This is a randomized study. Patients are stratified according to stage of disease (stage IIIB vs stage IV vs recurrent or progressive after surgery and/or radiotherapy), performance status (0-1 vs 2), and age (under 70 vs 70 and over). Patients are randomized to one of two treatment arms. Arm I receives paclitaxel IV over 3 hours on day 1 of each course. Arm II receives paclitaxel as in Arm I, followed by carboplatin IV over 1 hour. Treatment is repeated every 21 days for 6 courses in the absence of tumor progression or unacceptable toxicity. Quality of life assessments are conducted before treatment and at 2, 6, 9, and 12 months. Patients are followed every 3 months for 2 years, then every 6 months until disease progression or death.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically proven non-small cell lung cancer (adenocarcinoma, large cell, squamous cell, or mixture) Stage IIIB due to any of the following: Malignant pleural effusion Supraclavicular node involvement Contralateral hilar node involvement Not eligible for CALGB protocols of combined therapy and chest irradiation Stage IV Any stage that has recurred or progressed after surgery or radiotherapy Measurable or evaluable disease Does not include the following: Bone metastases Pleural or peritoneal effusions Irradiated lesions, unless progression documented after radiation therapy No CNS metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: CALGB 0-2 Life expectancy: Not specified Hematopoietic: Granulocyte count at least 1500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin less than 1.5 mg/dL SGOT less than 2 times the upper limit of normal (ULN) Renal: Creatinine no greater than 2 times ULN Other: No prior or concurrent malignancy except: Curatively treated carcinoma in situ of the cervix Curatively treated breast cancer Curatively treated basal cell or squamous cell skin cancer At least 5 years since any nonrecurrent primary tumor surgically resected without administration of adjuvant radiation therapy or chemotherapy HIV negative

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy No other concurrent chemotherapy Endocrine therapy: No concurrent hormones except steroids for adrenal failure, hormones for nondisease related conditions (e.g., insulin for diabetes), or dexamethasone Radiotherapy: At least 2 weeks since prior radiotherapy See Disease Characteristics Surgery: Prior surgery allowed See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 584 (Actual)
Dates: Start 1997-10; Primary Completion 2004-12 (Actual); Study Completion 2006-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rogerio Lilenbaum, MD, Study Chair — Yale University
Locations (35):
- United States (35):
  - University of California San Diego Cancer Center, La Jolla, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - University of Illinois at Chicago Health Sciences Center, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Marlene & Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Roswell Park Cancer Institute, Buffalo, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Presbyterian Hospital - Cornell Campus, New York, New York
  - Mount Sinai Medical Center, NY, New York, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center of Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Tennessee, Memphis Cancer Center, Memphis, Tennessee
  - Vermont Cancer Center, Burlington, Vermont
  - Massey Cancer Center, Richmond, Virginia
  - MBCCOP - Massey Cancer Center, Richmond, Virginia

REFERENCES:
- [Background] Lamont EB, Herndon JE 2nd, Weeks JC, Henderson IC, Lilenbaum R, Schilsky RL, Christakis NA; Cancer and Leukemia Group B. Measuring clinically significant chemotherapy-related toxicities using Medicare claims from Cancer and Leukemia Group B (CALGB) trial participants. Med Care. 2008 Mar;46(3):303-8. doi: 10.1097/MLR.0b013e31815cecc3. PMID 18388845
- [Background] Lamont EB, Herndon JE 2nd, Weeks JC, Henderson IC, Lilenbaum R, Schilsky RL, Christakis NA. Criterion validity of Medicare chemotherapy claims in Cancer and Leukemia Group B breast and lung cancer trial participants. J Natl Cancer Inst. 2005 Jul 20;97(14):1080-3. doi: 10.1093/jnci/dji189. PMID 16030306
- [Result] Lilenbaum RC, Herndon JE 2nd, List MA, Desch C, Watson DM, Miller AA, Graziano SL, Perry MC, Saville W, Chahinian P, Weeks JC, Holland JC, Green MR. Single-agent versus combination chemotherapy in advanced non-small-cell lung cancer: the cancer and leukemia group B (study 9730). J Clin Oncol. 2005 Jan 1;23(1):190-6. doi: 10.1200/JCO.2005.07.172. PMID 15625373
- [Result] Lilenbaum RC, Herndon J, List M, et al.: Single-agent (SA) versus combination chemotherapy (CC) in advanced non-small cell lung cancer (NSCLC): a CALGB randomized trial of efficacy, quality of life (QOL), and cost-effectiveness. [Abstract] Proceedings of the American Society of Clinical Oncology 21: A-2, 2002.